CLINICAL TRIAL: NCT01373424
Title: Natural History and Biospecimen Repository for Dystonia; Comprehensive Rating Tools for Cervical Dystonia; Validity & Reliability of Diagnostic Methods & Measures of Spasmodic Dysphonia
Brief Title: The Dystonia Coalition Natural History and Biospecimen Repository for Isolated Dystonias
Acronym: DCP
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Office of Rare Diseases (ORD) (NIH); Allergan (Industry); Dystonia Study Group (Other)
Responsible Party: Principal Investigator, Hyder A. Jinnah, MD, PhD, Principal Investigator, Emory University
Other Study IDs: IRB00046266; U54TR001456 (NIH); RDCRN#6301 (Other: Other); U54NS065701 (NIH)
Record Dates: First submitted 2011-06-02; First posted 2011-06-15 (Estimated); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Dystonia
Keywords: Observational study; Cross-sectional and Prospective study; Cohort and case-control study
MeSH Terms: conditions — Dystonia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole blood, DNA, white blood cells, cell lines
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Cervical dystonia: People diagnosed with cervical dystonia
- Laryngeal dystonia: People diagnosed with laryngeal dystonia
- Other voice disorders: People diagnosed with a voice disorder other than laryngeal dystonia - enrollment for this group is complete
- Craniofacial dystonia: People diagnosed with craniofacial dystonia (including blepharospasm, meige syndrome, and oromandibular dystonia)
- Limb dystonia: People diagnosed with limb dystonia
- All other isolated dystonias: People diagnosed with any isolated dystonia not listed in descriptions of other cohorts
- Myoclonus dystonia: People diagnosed with myoclonus dystonia
- Dopa-responsive dystonia: People diagnosed with dopa-responsive dystonia

SUMMARY:
Dystonia is a disorder characterized by excessive involuntary contraction of muscles with repetitive and patterned movements. The isolated dystonias are the most common type of dystonia and include Limb dystonias (like writer's cramp), Cervical dystonia (spasmodic torticollis), Laryngeal dystonias (like spasmodic dysphonia), and Craniofacial dystonias (like blepharospasm). The purpose of this study is to create resources to help learn more about the isolated dystonias, myoclonus dystonia, and dopa-responsive dystonia and to develop and validate various dystonia rating scales.

DETAILED DESCRIPTION:
This collaborative, international effort has one primary goal. This is to create a biospecimen repository and associated clinical database to be used as a resource for dystonia and related disease research. Across sites, the investigators hope to enroll at least 5,000 adult patients.

Subjects of this study will be asked to complete a neurological exam which will be video recorded, complete some questionnaires, and donate a blood sample. A study visit will take between 45 minutes and 1 hour. All subjects will be asked to return every 1, 2, 3, or 4 years for a one hour follow-up visit. People may participate in this study without agreeing to participate in the follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with isolated dystonia or myoclonus dystonia or dopa-responsive dystonia
* To be included in laryngeal dystonia group, nasolaryngoscopy (voice box exam) must have been completed to confirm diagnosis (this voice box exam is not part of the study)

Exclusion Criteria:

* Any evidence of a secondary cause for dystonia (other than myoclonus dystonia or dopa-responsive dystonia)
* Less than 2 months since last botulinum toxin injection
* Inability to provide informed consent
* Significant medical or neurological conditions that preclude completing the neurological exam
* Significant physical or other condition that would confound diagnosis or evaluation, other than dystonia or tremor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with dystonia are eligible to participate as long as they are above age 18 and fit the eligibility criteria. The coordinator at the site you contact can tell you more about this.
Sampling Method: Non-Probability Sample
Enrollment: 3265 (Actual)
Dates: Start 2011-01; Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Observational | 7 years
  There is no primary outcome measure as this is an observational study.

CONTACTS AND LOCATIONS:
Overall Officials: H. A. Jinnah, MD, PhD, Principal Investigator — Emory University
Locations (42):
- United States (34):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Mayo Clinic, Arizona, Scottsdale, Arizona
  - Parkinson's and Movement Disorders Institute, Fountain Valley, California
  - University of California, San Diego, La Jolla, California
  - University of Colorado, Denver, Denver, Colorado
  - University of Florida, Gainesville, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Rush University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - National Institutes of Health, Bethesda, Maryland
  - Parkinson's and Movement Disorders Center of Maryland, Elkridge, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Washington University in St. Louis, St Louis, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - Mount Sinai Beth Israel, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Wake Forest, Winston-Salem, North Carolina
  - Sanford Health - Fargo, Fargo, North Dakota
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pennsylvania, Parkinson's Disease and Movement Disorders Center, Philadelphia, Pennsylvania
  - University of Tennessee, Memphis, Tennessee
  - University of Texas, Southwestern, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Neurological Institute, Houston, Texas
  - University of Texas, Houston, Texas
  - James Madison University, Harrisonburg, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Booth Gardner Parkinson's Care Center, Kirkland, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Westmead Hospital, Westmead, Australia
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - Toronto Western Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
- Hopital de la Salpetriere, Paris, France
- University Hospital of Schleswig-Holstein, Lübeck, Germany
- University of Rome, Rome, Italy
- University College London Institute of Neurology, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data is available to researchers with appropriate ethics board approvals. Researchers may contact the Dystonia Coalition PI or coordinator at Emory University or the RDCRN Data Management and Coordination Center for more information.

REFERENCES:
- [Derived] Patel N, Hanfelt J, Marsh L, Jankovic J; members of the Dystonia Coalition. Alleviating manoeuvres (sensory tricks) in cervical dystonia. J Neurol Neurosurg Psychiatry. 2014 Aug;85(8):882-4. doi: 10.1136/jnnp-2013-307316. Epub 2014 May 14. PMID 24828895
- See also: Dystonia Coalition website — http://rdcrn.org/Dystonia

DOCUMENTS (1):
  • Informed Consent Form (2016-08-03): https://cdn.clinicaltrials.gov/large-docs/24/NCT01373424/ICF_000.pdf